CLINICAL TRIAL: NCT00822289
Title: Effect of Radioactive Iodine on Eradication of Helicobacter Pylori in Patients Treated for Thyroid Diseases
Brief Title: The Effect of Radioactive Iodine Administration for Thyroid Diseases on H.Pylori Eradication
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Rabin Medical Center (Other)
Responsible Party: Haim Shmuely, MD, Rabin Medical Center
Other Study IDs: 5071
Record Dates: First submitted 2009-01-13; First posted 2009-01-14 (Estimated); Last update posted 2009-01-14 (Estimated); Status verified 2009-01

CONDITIONS: Helicobacter Pylori Infected Patients; Thyroid Cancer Patients; Hyperthyroidism
Keywords: radioactive iodine; Helicobacter pylori; Thyroid diseases; CagA
MeSH Terms: conditions — Hyperthyroidism; Thyroid Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Because of the high iodine uptake in the stomach, radioactive iodine treatment for thyroid diseases (cancer or hyperthyroidism) or radioactive iodine administered for thyroid scan may be able to eradicate H.pylori infection from the stomach of patients infected with H.pylori.

Also to test the hypothesis that CagA virulent strains of H.pylori are more common in patients with thyroid cancer than with other thyroid diseases.

DETAILED DESCRIPTION:
Objective To test eradicate H.pylori after administration of radioactive iodine (131I) to patients with thyroid diseases and to evaluate their H.pylori CagA status .

Design Observational study

Setting

The Isotopic Institute at the Rabin Medical Center, Campus Beilinson Patients Consecutive patients with thyroid diseases referred to the Isotopic Institute at the Rabin Medical Center, Campus Beilinson for either radioactive iodine (131I) thyroid scan or radioactive iodine (131I)treatment for their disease, will be screened, prior to the radioactive iodine, for H. pylori infection and CagA protein by serology. Patient with positive serology for H. pylori will be tested for active gastric infection using the H.pylori stool antigen test. The study population will include all patients who tested positive for H.pylori both by serology and stool antigen tests. Six to eight weeks and 6 month after administration of radioactive iodine (131I) treatment , stool antigen or H.pylori will be tested again to confirm persistence of H.pylori eradication.

Main Outcome Measure confirmed H.pylori eradication by the stool antigen test. The rate of infection with virulent and caricogenic CagA H.pylori ,will be tested using the immunoblot assay.

Summary

We will test in this study whether Helicobacter pylori is eradicated, after radioactive iodine (131I) administration, from the stomach of patients with thyroid diseases. The rate of CagA virulent and carcinogenic H.pylori infection in theses patients will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients between the ages of 18 and 80.
* Patients with diagnosed thyroid disease referred for thyroid scan or treatment with radioactive iodine (131I).
* Patients who provide informed consent

Exclusion Criteria:

* Patients without diagnosed thyroid disease.
* Patients who are pregnant or breast feeding.
* Patients who have received previous treatment for H. pylori infection.
* Patients taking proton pump inhibitors.
* Patients with recent or current use of antibiotics.
* Patients allergic to iodine (131I).

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with thyroid diseases referred to the Isotopic Institute at the Rabin Medical Center, Campus Beilinson for either radioactive iodine (131I) thyroid scan or radioactive iodine (131I)treatment for their disease, will be tested, prior to the radioactive iodine, for H. pylori infection and CagA protein by serology. Patient with positive serology for H. pylori will be tested for active gastric infection using the H.pylori stool antigen test. The study population will include all patients who tested positive for H.pylori both on serology and stool antigen tests. Six to eight weeks and 6 month after administration of radioactive iodine (131I) , stool antigen or H.pylori will be tested again to confirm persistence of H.pylori eradication.
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2009-02

SECONDARY OUTCOMES:
To determine whether CagA helicobacter pylori infection is more prevalent in patients with thyroid diseases compared to other thyroid diseases | 2 years